CLINICAL TRIAL: NCT01653340
Title: A Feasibility Clinical Trial to Evaluate High Frequency Spinal Cord Stimulation for the Treatment of Patients With Chronic Migraine
Acronym: rCM HF-SCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Paolo Martelletti, Professor, Internal Medicine, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE100112; 2012-002005-22 (EudraCT Number)
Record Dates: First submitted 2012-07-24; First posted 2012-07-31 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Refractory Chronic Migraine
Keywords: Refractory Chronic Migraine; Medically Intractable Chronic Migraine; High Frequency Spinal Cord Stimulator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High Frequency Spinal Cord Stimulation through Senza™ (Experimental): During the trial implant of Senza™, High Frequency Spinal Cord Stimulator for Refractory Chronic Migraine, the 2 leads will be positioned to cover the C2-C3 cervical levels.
  Over the following 2 weeks, the investigator will optimize therapy delivery by identifying the stimulation settings providing maximal headache pain relief.
  The subject will be asked to attend the clinic at the end of the trial period. Together with his/her physician, the subject will discuss his/her experience over the past 2 weeks (satisfaction with the therapy), and decide whether or not move forward with a Nevro Senza IPG.
  The Nevro Senza IPG will be implanted in the buttock or abdomen area as outlined in the Physician's Manual. Fluoroscopy and impedance measurements may be used during the procedure to confirm lead placement and location.
  Before hospital discharge, the IPG will be programmed with the optimal settings identified during the trial phase.
  Interventions: Device: Senza™, High Frequency Spinal Cord Stimulator for Refractory Chronic Migraine

INTERVENTIONS:
Device: Senza™, High Frequency Spinal Cord Stimulator for Refractory Chronic Migraine — http://nevro.com/corporate/system-us

SUMMARY:
The purpose of this study is to assess short- and long-term safety, tolerability and efficacy of cervical High Frequency Spinal Cord Stimulation (HF-SCS) in patients suffering from chronic migraine refractory to conventional medical therapy.

DETAILED DESCRIPTION:
1. Introduction 1.1 Background Migraine is a common disabling headache disorder. Patients with Chronic Migraine (CM) experience headache on a minimum of 15 days per month. CM is associated with significant disability and reduced quality of life .

   Since the late 1990s, there has been considerable progress in neurostimulation techniques to treat medically intractable chronic-headache syndromes patients, by applying peripheral-nerve stimulation to patients . It is indeed well demonstrated that a non-painful stimulation of peripheral nerves can elicit analgesic effects, and that occipital nerve stimulation (ONS), by retrograde activation of the trigemino-cervical complex can provide effective pain relief in patients with headache disorders, including migraine. Recently, high cervical spinal cord stimulation (SCS) has been tested for the treatment of chronic cluster headache , highlighting a potential benefit of SCS over ONS: SCS exerts an immediate and almost maximal effect, which allows a test phase prior to implantation of the pulse generator with the possibility of removing the electrode in case of insufficient pain relief.

   Both SCS and ONS produce paresthesia, an unpleasant tingling sensation for the patients In recent prospective studies, a new modality of SCS, High Frequency (HF) SCS, has been demonstrated to be effective and safe in a chronic pain population, the Failed Back Surgery Syndrome (FBSS) population . High Frequency SCS differs from conventional SCS in several ways, which present significant advantages to both the patients and the healthcare professionals: 1) absence of paresthesia (tingling) which leads to greater patient comfort and acceptance of the therapy, 2) shorter procedural time as no paresthesia mapping is needed, and 3) increased efficacy compared to conventional SCS, demonstrated in the FBSS population. Additionally, HF SCS has a similar safety profile as conventional SCS.

   HF-SCS may thus combine the advantage of paresthesia free therapy (and thus greater patient tolerability of the therapy) with the possibility of testing the therapy during a trial phase prior to the implantation of a permanent pulse generator.
2. Study Objective, Outcomes, and Design 2.1 Objective The objective of this study is to investigate the safety, efficacy and tolerability of high frequency (HF) Spinal cord stimulation (SCS) for the treatment of patients with chronic migraine.

   2.2 Outcomes
   * Change of frequency in headache days from baseline;
   * Change of frequency in migraine days from baseline;
   * Change in frequency of moderate/severe headache days from baseline;
   * Change in headache pain Visual Analog Scale (VAS) score from baseline;
   * Change in HIT-6 score from baseline;
   * Change in Migraine Disability Assessment (MIDAS) Score from baseline;
   * Change in frequency of triptans intake from baseline;
   * Patient Global Impression of Change (PGIC);
   * Change in Quality of Life from baseline;
   * Change in the number of sleep disturbances per night from baseline;
   * Incidence of device-related adverse events.

   2.3 Target Size This feasibility study will enroll a minimum of 10 subjects and a maximum of 20 subjects.

   Each subject will undergo a trial phase of the therapy. If the trial is successful, the subjects will be followed-up for 6 months, with regular clinic follow-up visits.

   It is expected that the first subject will be enrolled in June 2012. The last subject is expected to complete the study follow-up period by January 2013.

   2.4 Devices Used

   The Senza™ System, manufacturer by Nevro (Menlo Park, USA), received CE mark in 2010 for use as an aid in the management of chronic intractable pain of the lower trunk and/or limbs. The Senza System is similar to other available SCS systems in design and function. However, Nevro's proprietary waveform algorithms may eliminate unwanted side effects, improve subject experience and potentially provide better pain relief.

   Similar to the commercial systems, the Senza System includes lead(s), anchor(s), extension(s), trial stimulator, implantable pulse generator (IPG), charger, patient remote control, and clinician programmer. Additional components include surgical tools, cables and various other accessories for use in the placement of the leads and IPG.
3. Selection and Withdrawal of Subjects

   This study will recruit subjects with chronic headache migraine as per the International Classification of Headache Disorders (2nd edition) .

   3.1 Inclusion/Exclusion Criteria

   To participate in the study, the subject must meet all of the following criteria:

   Include a subject who has (is):
   * An adult between the age of 18 and 65
   * Capable of providing informed consent
   * A diagnosis of chronic (>15 or more headache-days per 4 week period for more than 3 months, with an headache-day being defined as a day with an attack lasting a minimum of 4 hours) migraine refractory to conventional medical treatment (has failed at least 2 preventive and 2 abortive drugs) as per the ICHD-II guidelines.
   * On optimal and stable preventive headache pharmacological migraine therapy for at least 2 months
   * Failed treatment with Onabotulinumtoxin A for 12 months
   * Able to comply with the requirements of the study visits and self-assessment questionnaires Able to provide informed consent and willing to comply with study procedures

   Exclude a subject who has (is):
   * medication-overuse headache
   * Had treatment with Onabotulinumtoxin A in the last 3 months
   * An already implanted active medical device
   * A contraindication to the cervical placement of SCS lead
   * A life expectancy of less than 1 year
   * A female of child bearing potential who is pregnant/lactating or not using adequate birth control
   * Beck Depression Inventory score of >24
   * Evidence of an active disruptive psychological/psychiatric disorder or other known condition significant enough to impact perception of pain (e.g. fibromyalgia), compliance of intervention and/or ability to evaluate treatment outcome as determined by the Investigator
   * Addiction to any of the following: illicit drugs, alcohol (5 or more drinks/day), and/or medication
   * Bleeding diathesis such as coagulopathy or thrombocytopenia
   * Immuno-compromised and at risk for infection
   * Diabetic which is not under control as determined by the Investigator
   * Unresolved issue of secondary gain
   * Inability to manage the technical demands of the SCS equipment
   * Currently participating in a randomized clinical trial with an active treatment arm or planned to be enrolled in another clinical trial 3.2 Subject Early Withdrawal

   A subject may be withdrawn early from the study for the following reasons:
   * Adverse event
   * Non-compliance
   * At the discretion of the Investigator
   * Subject withdrawal of consent
   * Study is stopped by the Investigator or Ethics Committee (EC) 3.3 Device Explantation At the discretion of the Investigator or subject, the IPG and/or the leads(s) may be explanted from a subject. If the explantation is as a result of an unanticipated adverse device effect (UADE) or device failure, the Investigator will send the explanted devices and accessories (i.e., Remote Control) to Nevro for device analysis.

   If the subject is experiencing an adverse event related to the explant, the subject will be followed until resolution of that adverse event or determination that the subject's condition is stable. The Investigators or the EC may suspend or terminate the study early at any time. If the study is suspended or terminated prematurely, all currently enrolled subjects will be withdrawn from the study.
4. Treatment of Subjects/Study Procedures 4.1 Screening/enrollment The Investigator will identify potential study candidates who are likely to meet study inclusion and exclusion criteria and discuss participation in the study. If the subject agrees, the Investigator and research staff will meet with the subject to review details of the study. The subject will have the opportunity to read the informed consent and ask any questions. This study is entirely voluntary. Subject consent will be obtained in accordance and in compliance with Good Clinical Practice guidelines and Italian regulations.

   If the subject agrees to participate in the trial he/she will sign the consent form. After the subject provides informed consent, he/she is considered enrolled into the study.

   The subject will be asked to attend the clinic to complete a series of subject questionnaires to gather information on their condition and current level of pain, disability and affected lifestyle metrics.

   Enrolled subjects will undergo a 2 week HF-SCS trial. 4.2 Trial Phase During the trial implant, the 2 leads will be positioned to cover the C2-C3 cervical levels.

   Over the following 2 weeks, the investigator will optimize therapy delivery by identifying the stimulation settings providing maximal headache pain relief.

   During this period, the patient will complete daily a headache diary to record their headache frequency, intensity and duration.

   The subject will be asked to attend the clinic at the end of the trial period. Together with his/her physician, the subject will discuss his/her experience over the past 2 weeks (satisfaction with the therapy), and decide whether or not move forward with a Nevro Senza™ IPG. If the subject chooses not to move ahead, she/he will be given alternative treatment options by the physician, and no further follow up study procedures will be required.

   During the trial phase, and until the 3 month follow-up visit, the physician will try to keep the headache medication as stable as possible, in order to avoid confounding factors when investigating the efficacy of the therapy Permanent Implant The Nevro Senza™ IPG will be implanted in the buttock or abdomen area as outlined in the Physician's Manual. Fluoroscopy and impedance measurements may be used during the procedure to confirm lead placement and location.

   As per the Investigator's standard clinical practice the subject will be placed on prophylactic antibiotics as a preventative for skin flora (bacteria) infections. Subjects will follow the Investigator's protocol for anticoagulant therapy and other medications.

   Before hospital discharge, the IPG will be programmed with the optimal settings identified during the trial phase. The Patient Manual will be reviewed with the subject and a copy will be given to the subject for future reference 4.3 Follow-Up Visits Subjects implanted with an IPG will be asked to attend in-clinic visits at 3 and 6 months post IPG implantation.

   During these visits, the subjects will undergo a clinical assessment and the following data will be collected on Case Report Forms (CRFs):
   * Medication usage
   * Headache Impact Test (HIT)-6 questionnaire
   * Migraine Disability Assessment (MIDAS) questionnaire
   * Quality of Life questionnaire
   * Patient Global Impression of Change (PGIC) scale
   * Patient Sleep disturbances

   The patient headache diary will be reviewed and a new one provided for the next follow-up period.

   During these visits, all Adverse Events will be documented. Until the 3 month follow-up visit, the physician will try to keep the headache medication as stable as possible, in order to avoid confounding factors when investigating the efficacy of the therapy

   At the end of the 6-months period, the study will be completed and the subjects will continue to be followed-up as per the center standard practice.

   4.4 Interim/Unscheduled Visits Subjects may be seen in the clinic for interim/unscheduled visits at any time during study. Possible reasons for an interim/unscheduled visit include the need to modify device programming to adjust pain relief, or for an adverse event. Such visits will be documented on CRFs.
5. Data Measures and Analysis Both qualitative and quantitative data will be collected and analysed. Table 1: Data Collection per visit

   CRFs Enrollment Trial implant End of trial IPG implant Month 3 Month 6 Enrollment x Medical history x Medication usage x x x x Questionnaires (HIT-6, MIDAS, QoL, PGIC) x x x x Implant details x x Patient diary x x x x x Adverse Event x x x x x

   General descriptive measures will include counts and percentages for categorical measures and the mean, standard deviation, median, and minimum and maximum values for continuous data.

   Non-parametric 2-tailed cross sectional and pair-wise comparisons will be undertaken. Simple linear and non-linear regression will be used to calculate predictor values from the vertebral level data collected. Significance will be set at the 0.05 level.

   Additional analyses may be conducted.
6. Adverse Events 6.1 Definitions The definitions presented in this section allow for a clear understanding of adverse event data collection and reporting requirements.

   6.1.1 Adverse event An adverse event (AE) is defined as any undesirable clinical occurrence in a subject that appears or worsens in the clinical study (as compared to the subject's baseline health) and is any untoward medical occurrence defined as an unintended disease or injury or untoward clinical signs (including abnormal laboratory findings) in a subject whether or not related to the investigational or commercial medical device. This definition includes events related to the study medical devices and events related to the study procedures. An AE is also any event related to any underlying medical condition, present at baseline, which increases in severity by a clinically meaningful amount during the study as determined by the Investigator.

   Adverse events will be summarized by type, severity, treatment/intervention provided, relationship to the device/procedure, and resolution.

   As the primary efficacy measure in this study is pain, back and leg pain does not need to be reported as an adverse event unless it meets the definition of a serious adverse event. However, Investigators may, at their discretion, report any pain-related adverse events during the study.

   Pre-existing conditions will not be reported as an adverse event unless there has been a substantial increase in the severity or frequency of the problem which has not been attributed to natural history.

   6.1.2 Serious adverse events

   A serious adverse event is an adverse event that:
   * Leads to death
   * Leads to a serious deterioration in the health of the subject that:
   * Results in life-threatening illness or injury
   * Results in a permanent impairment of a body structure or a body function
   * Requires in-subject hospitalization or prolongation of existing hospitalization
   * Results in medical or surgical intervention to prevent permanent impairment to body structure or a body function
   * Leads to fetal distress, fetal death, or a congenital abnormality or birth defect 6.1.3 Adverse device effect

   An adverse device effect (also called a device-related adverse event) is an adverse event with a reasonable possibility that the device caused or contributed to the event. During this clinical investigation an event should be considered related to the device when it is the result of:
   * The device components (e.g., lead, extension, IPG)
   * The implant procedure
   * The therapy/stimulation 6.1.4 Serious adverse device effect An untoward medical occurrence that happens in a subject, is related to the investigational device, procedure, or therapy and is serious, but is not unanticipated is a serious adverse device effect (SADE). Untoward medical occurrences that are anticipated, i.e. are unsurprising, are identified in the investigator's brochure or protocol and informed consent form.

   Anticipated adverse events related to the device, procedure or therapy are listed in section 7, Risk/Benefit.

   6.1.5 Unanticipated serious adverse device effect An untoward medical occurrence that happens in a subject, is related to the investigational device, device procedure, or therapy, is serious, and is unanticipated is classified as an unanticipated serious adverse device effect (USADE).

   Anticipated adverse events related to the device, procedure or therapy are listed in Section 7, Risk/Benefit.

   6.1.6 Severity

   The Investigator will use the following definitions to rate the severity of each adverse event:
   * Mild: Awareness of a sign or symptom that does not interfere with the subject's usual activity or is transient, resolved without treatment and no sequelae
   * Moderate: Interferes with the subject's usual activity or requires symptomatic treatment
   * Severe: Symptom(s) causing severe discomfort with significant impact of the subject's usual activity and requires treatment 6.2 Reporting The Investigator will assess the subject for adverse events and capture the required adverse event information in the subject records or an appropriate study form. Adverse events can be based on subject report. Subjects should be instructed to contact their physician in the case of emergency, as described in the informed consent.

   All AEs will be followed until the event is resolved (with or without sequelae). If an event is ongoing at the time study completion of termination, the subject will be followed until resolution or Investigator determination that the subject's condition is stable.

   The Investigator is responsible for reporting information regarding specific AEs (e.g. SAEs and UADEs) to the appropriate EC as required by local regulations. The Investigator will also report any UADEs and appropriate device related AEs to Nevro.
7. Risk/Benefit 7.1 Potential Risks A risk analysis was completed by Nevro Corporation in accordance with ISO 14971 - Application of Risk Management for Medical Devices. This analysis showed that the Senza System exhibits a safety profile equivalent to the commercially available stimulators.

   In an effort to report all of the potential risks for this study, all adverse events attributed to the device, procedure or stimulation therapy reported in a review of key SCS literature (Cameron 2004; Kumar et al. 2007) are described in this section. Table 2 lists the adverse events that were reported in these articles in order of frequency reported in the Cameron article. These are foreseeable risks that are presented in the informed consent and are typical of commercial SCS systems.

   Other adverse events which may potentially occur, but were not reported in the Cameron and Kumar articles, include: increased intensity, duration, or frequency or back and/or leg pain, uncomfortable stimulation of tissue around the leads including skin and muscle, development of pain symptoms in a new location, thrombosis, nerve injury, seizure, and death.

   As the primary efficacy measure in this study is pain, headache pain does not need to be reported as an adverse event unless it meets the definition of a serious adverse event. However, Investigators may, at their discretion, report any pain-related adverse events.

   Table 2: Risks Associated with Spinal Cord Stimulation Cameron 2004 Kumar 2007 n = 2107-2972

   % n = 84

   % Lead migration 13.2 9.5 Lead breakage 9.1 2.4b Infection 3.4 8.3a Hardware malfunction 2.9 nr Unwanted stimulation 2.4 1.2c Battery failure 1.6 nr Other 1.4 nr Pain over implant 0.9 6.0 Loose connection 0.4 1.2 CSF leak 0.3 1.2d Hematoma 0.3 nr Skin erosion 0.2 nr Allergic reaction 0.1 nr Paralysis 0.03 nr Neurostimulator pocket fluid collection/seroma 0.0 4.8 Intermittent stimulation 0.0 nr Epidural hemorrhage 0.0 nr Loss of therapeutic effect, loss of paresthesia, or unpleasant paresthesia nr 7.1 Techniquee nr 2.4 IPG migration nr 1.2 Abbreviations: nr, not reported. a reported as "infection and wound breakdown" b reported as "lead extension fracture/torqued contacts" c reported as "anteriorly placed electrode caused shocks" d reported as "dural tear" e cap not installed on IPG when only one lead was implanted (1), lead cut during implant (1)

   7.2 Possible Benefits The Senza System has received CE mark approval for use in the treatment of chronic intractable pain. The hazards and mitigation mechanisms were identified and risk factors were calculated for each of the identified hazards and were found to be within the acceptance criterion. The results of the risk analysis concluded that the benefit of providing pain relief for subjects suffering from chronic intractable pain outweighs the residual risks that may be posed by the use of this device.

   The desired benefit is the improvement in the status of the patient's refractory pain. There is however, no guarantee that this will happen. Results of prior and on-going clinical studies show that the Senza System offers an opportunity for improved pain relief in this chronic intractable pain population. Thus, by participating in this study the information gathered will add to the understanding of treatment options for patients with chronic migraine. This knowledge may advance medical science and may benefit other patients with chronic pain and potentially society at large.
8. Conduct of Study

   8.1 Statement of Study Compliance The study will be performed in accordance with ISO 14155-2011, Good Clinical Practice (GCP) guidelines, recommendations guiding physicians in biomedical research involving humans adopted by the 18th World Medical Assembly, Helsinki, Finland (1964 and later revisions). The Investigator, as required by the local regulations should notify the EC in writing after completion, termination, or discontinuation of the study at the site. If study is discontinued due to safety concerns, the Investigator will notify the EC immediately.

   8.2 Investigator Responsibilities The Investigator is responsible for ensuring that the investigation is conducted according to the study protocol, and applicable ISO EN 14155-2011, data protection regulations, and any other applicable Ethics Committee= requirements.

   The Investigator(s) shall be responsible for the day-to-day conduct of the investigation as well as for the safety and well-being of the human patients involved in the clinical investigation.

   It is the responsibility of the Investigator to obtain approval of the study protocol from the EC and to keep the EC informed of any serious adverse events, unanticipated adverse device effects, and amendments to the protocol. All correspondence with the EC should be filed by the Investigator.

   8.3 Quality Control and Quality Assurance All documents and data shall be produced and maintained in such a way to assure control of documents and data to protect the patient's privacy as far as reasonably practicable. Representatives of the applicable regulatory authorities are permitted to inspect the study documents (e.g., study protocol, CRFs, and original study-relevant medical records/files) as needed. All attempts will be made to preserve patient confidentiality.

   8.4 Ethics The Investigator is a physician whose first responsibility is to the care of the patient. Should individual care conflict with study requirements, it is understood that the care of the patient is foremost. In all respects, this study shall be conducted pursuant to the "Declaration of Helsinki: Recommendations Guiding Medical Doctors in Biomedical Research Involving Human Subjects".

   At all times, the Investigators are to follow this confirmatory study plan, abide by all Good Clinical Practice requirements set by prevailing national law and any EC regulations.

   8.5 Termination or Suspension of the Investigation The study may be terminated when all of the requirements of the protocol have been fulfilled. Patients will be considered to have completed all study requirements following completion of the 6 month visit.

   The Investigators or EC may suspend or terminate the study early at any time. If the study is suspended or terminated prematurely, all currently enrolled patients will be withdrawn from the study. If there is an ongoing event related to the device or therapy, the patient will be followed until resolution of that adverse event or determination that the subject's condition is stable.
9. Data Handling and Recordkeeping

All documents will be maintained by the Investigator. The data will be collected using appropriate questionnaires and will be secured by the Investigator. The Investigator will be required to keep study records as dictated by local regulations.

Appendix A - Responsibilities of Investigators

The Investigator is responsible for ensuring that this clinical study is conducted according to all conditions of the HREC approval and applicable regulations. The Investigator is responsible for ensuring that informed consent is obtained from all subjects prior to any diagnostic tests or treatments that are outside the standard course of treatment that would be followed if this subject were not being considered for enrollment in this clinical study.

Subjects will be informed that they are free to refuse to participate in this clinical study without loss of benefits to which they are otherwise entitled, and that if they choose to participate, they may withdraw at any time without prejudice to future care. The informed consent approved by the HREC must be signed prior to study participation. The original signed informed consent for each subject must be retained by the Sponsor Investigator.

Other specific responsibilities of the Sponsor Investigator include:

Awaiting Approval The Investigator may discuss with a subject their interest in participating in the clinical study, but shall not request the written informed consent nor allow any subject to participate in the clinical study before HREC and other necessary approvals are received.

Subject records Subject records include signed informed consent forms, copies of all completed case report forms and supporting documents (laboratory reports, reports of diagnostic tests, medical records, etc.) and records of exposure of each subject to the device. Informed consent must comply with EN/ISO 14155-2011.

Documentation of the Use of the Device without Informed Consent The Investigator must document use of the device without Informed Consent. The Investigator is responsible for reporting device usage without prior informed consent per the applicable regulations.

Unanticipated Adverse Device Effects The Investigator is responsible for maintaining records of all reports and information pertaining to unanticipated adverse device effects.

Ethics Committee Information The Investigator is responsible for maintaining all information pertaining to EC review and approval of this clinical study including a copy of the EC letter approving the clinical study, a blank informed consent form approved by the EC and that the EC approved the protocol.

ELIGIBILITY:
Inclusion Criteria:

* An adult between the age of 18 and 65

  * Capable of providing informed consent
  * A diagnosis of chronic (>15 or more headache-days per 4 week period for more than 3 months, with an headache-day being defined as a day with an attack lasting a minimum of 4 hours) migraine refractory to conventional medical treatment (has failed at least 2 preventive and 2 abortive drugs) as per the ICHD-II guidelines.
  * On optimal and stable preventive headache pharmacological migraine therapy for at least 2 months
  * Failed treatment with Onabotulinumtoxin A for 12 months
  * Able to comply with the requirements of the study visits and self-assessment questionnaires Able to provide informed consent and willing to comply with study procedures

Exclusion Criteria:

* • medication-overuse headache

  * Had treatment with Onabotulinumtoxin A in the last 3 months
  * An already implanted active medical device
  * A contraindication to the cervical placement of SCS lead
  * A life expectancy of less than 1 year
  * A female of child bearing potential who is pregnant/lactating or not using adequate birth control
  * Beck Depression Inventory score of >24
  * Evidence of an active disruptive psychological/psychiatric disorder or other known condition significant enough to impact perception of pain (e.g. fibromyalgia), compliance of intervention and/or ability to evaluate treatment outcome as determined by the Investigator
  * Addiction to any of the following: illicit drugs, alcohol (5 or more drinks/day), and/or medication
  * Bleeding diathesis such as coagulopathy or thrombocytopenia
  * Immuno-compromised and at risk for infection
  * Diabetic which is not under control as determined by the Investigator
  * Unresolved issue of secondary gain
  * Inability to manage the technical demands of the SCS equipment
  * Currently participating in a randomized clinical trial with an active treatment arm or planned to be enrolled in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Frequency in headache days | three and six months
  Change of frequency in headache days from baseline
Frequency in migraine days | three and six months
  Change of frequency in migraine days from baseline
Frequency of moderate/severe headache days | three and six months
  Change in frequency of moderate/severe headache days from baseline

SECONDARY OUTCOMES:
headache pain Visual Analog Scale (VAS) | three and six months
  Change in headache pain Visual Analog Scale (VAS) score from baseline
HIT-6 | three and six months
  Change in HIT-6 score from baseline
Migraine Disability Assessment (MIDAS) | three and six months
  Change in Migraine Disability Assessment (MIDAS) Score from baseline
Frequency of triptans intake | three and six months
  Change in frequency of triptans intake from baseline
Patient Global Impression of Change (PGIC) | three and six months
  Patient Global Impression of Change (PGIC)
Quality of Life | three and six months
  Change in Quality of Life from baseline
sleep disturbances | three and six months
  Change in the number of sleep disturbances per night from baseline
Device-related adverse events | Three and six months
  Incidence of device-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Martelletti, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sant'Andrea Hospital, Roma, RM, Italy